CLINICAL TRIAL: NCT05627921
Title: The Effect of Botulinum Toxin and ESWT Applications on Spasticity and Functionality in Cerebral Palsy Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09.2022.1312
Record Dates: First submitted 2022-11-16; First posted 2022-11-28 (Actual); Last update posted 2022-11-28 (Actual); Status verified 2022-11

CONDITIONS: Cerebral Palsy, Spastic
Keywords: botilinum toxin; spasticity; eswt
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into two equal groups using the closed envelope system. The patients in the first group will be injected with Botulinum Toxin-A with the Stumplex device into the spastic muscle.
  The patients in the second group will be injected with Botulinum toxin with the same procedure. 1 week after the injection, patients will receive 3 sessions of radial ESWT treatment, 1 session/week. rESWT application will be applied with the 'MODUS ESWT' device and a 35 mm radial soft applicator will be used.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The person performing the examinations and evaluating the data was blind to the treatment administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- botulinum toxin group (Experimental)
  Interventions: Drug: Botilinum Toxin injection
- botilinum toxin and ESWT group (Experimental)
  Interventions: Device: Extracorporeal Shock Wave Therapy; Drug: Botilinum Toxin injection

INTERVENTIONS:
Device: Extracorporeal Shock Wave Therapy — Spastic muscles will be determined by examination. Botulinum toxin-A will be injected into the spastic muscles with Stumplex. 1 week after the injection, patients will receive 3 sessions of radial ESWT treatment, 1 session/week. rESWT application will be applied with the 'MODUS ESWT' device and a 35 mm radial soft applicator will be used. rESWT will be applied with a soft applicator. The soft applicator is designed for application to sensitive and painful areas and applications will be painless.Shock waves will be applied at 1500/beat, 8 Hz, 0.030 Mj/mm2, 2 bar per muscle.
  Arms: botilinum toxin and ESWT group
Drug: Botilinum Toxin injection — Spastic muscles will be determined by examination. Botulinum toxin-A will be injected into the spastic muscles with Stumplex.

SUMMARY:
Cerebral Palsy (CP) is a group of movement and posture disorders associated with a non-progressive affect during brain development that can cause limitation of activity and disability. The most common movement disorders in CP are spasticity and dystonia. Currently, the treatment of muscle stiffness called spasticity includes physiotherapy, casting and device, various drugs and surgical treatment. Botulinum toxin injection into the muscle also acts by reducing muscle contraction. ESWT is a method used in various musculoskeletal diseases. It has been previously applied to pediatric patients and has been shown to be effective and painless in ankle muscle stiffness. However, there are few studies investigating the effect of ESWT on functionality.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a permanent, non-progressive disorder in movement, posture, and motor development that occurs in the immature fetal or neonatal brain. Motor disturbances may be accompanied by secondary musculoskeletal problems such as spasticity and contractures. In the treatment of spasticity, various treatments such as exercise, occupational therapies, ultrasound, electrical stimulation, physiotherapy applications such as ESWT, orthoses, oral antispasticity agents, botulinum toxin injection, intrathecal baclofen, and surgery are applied. Botulinum toxin type A is one of the most widely used pharmacological treatments in the treatment of focal spasticity. Repeated injections may lead to the formation of neutralizing antibodies, resulting in a decrease in BoNT-A activity. In addition, a decrease in Botulinum toxin response may be observed due to the increase in intramuscular fat and connective tissue. In addition, in some patients with diffuse spasticity, the total dose of BoNT-A required may exceed the maximum dose. Therefore, various non-pharmacological treatment methods are recommended in addition to BoNT-A in the management of spasticity. Extracorporeal shock wave therapy (ESWT) is a treatment method for applying high pressure waves to the body. The effectiveness of ESWT on spasticity in patients with upper motor neuron damage has been demonstrated in previous studies. However, there are few studies investigating the effect of ESWT after BoNT-A injection on muscle tone, functionality and quality of life. Previous studies have shared the results of short-term follow-up after ESWT and BoNT-A injection.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of Spastic Cerebral Palsy confirmed by a pediatric neurologist, Patients with a spasticity value of at least 2 in the evaluation with the Modified Ashworth Scale (MAS), Patients with Botulinum Toxin injection indication by their physician, Having a mental level to understand the commands of the person making the assessment, agree to participate in the study

Exclusion Criteria:

* Patients diagnosed with dyskinetic, ataxic, mixed type cerebral palsy, Hypersensitivity to Onabotulinumtoxin A or any of the excipients, Infection at the planned injection site or sites, Having an uncontrolled epileptic seizure, Upper/lower extremity contracture, coagulopathy, Refusing to participate in the study, The patient is not oriented and cooperative, Contraindication of anesthesia for the group requiring anesthesia

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-07-15 (Estimated); Study Completion 2023-07-15 (Estimated)

PRIMARY OUTCOMES:
Modified Tardieu Scale | T0:Patients will be evaluated before botulinum toxin injection.
  The intensity of muscle tone is evaluated at different determined rates. At the joint, the first angle at which the increase in resistance is detected is recorded. The range of motion is compared to the angle at completion.
Modified Tardieu Scale | T1:Patients will be evaluated 1 week after botulinum toxin injection.
  The intensity of muscle tone is evaluated at different determined rates. At the joint, the first angle at which the increase in resistance is detected is recorded. The range of motion is compared to the angle at completion.
Modified Tardieu Scale | T2:Patients will be evaluated 1 month after botulinum toxin injection.
  The intensity of muscle tone is evaluated at different determined rates. At the joint, the first angle at which the increase in resistance is detected is recorded. The range of motion is compared to the angle at completion.
Modified Tardieu Scale | T3:Patients will be evaluated 3 months after botulinum toxin injection.
  The intensity of muscle tone is evaluated at different determined rates. At the joint, the first angle at which the increase in resistance is detected is recorded. The range of motion is compared to the angle at completion.
Modified Tardieu Scale | T4:Patients will be evaluated 6 months after botulinum toxin injection.
  The intensity of muscle tone is evaluated at different determined rates. At the joint, the first angle at which the increase in resistance is detected is recorded. The range of motion is compared to the angle at completion.

SECONDARY OUTCOMES:
Modified Ashworth Scale | T0:Patients will be evaluated before botulinum toxin injection.
  muscle tone 0 (0) - No increase in muscle tone 1 (1) - Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension
  1+ (2) - Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM 2 (3) - More marked increase in muscle tone through most of the ROM, but affect part(s) easily moved 3 (4) - Considerable increase in muscle tone passive, movement difficult 4 (5) - Affected part(s) rigid in flexion or extension
Modified Ashworth Scale | T1:Patients will be evaluated 1 week after botulinum toxin injection.
  muscle tone 0 (0) - No increase in muscle tone 1 (1) - Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension
  1+ (2) - Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM 2 (3) - More marked increase in muscle tone through most of the ROM, but affect part(s) easily moved 3 (4) - Considerable increase in muscle tone passive, movement difficult 4 (5) - Affected part(s) rigid in flexion or extension
Modified Ashworth Scale | T2:Patients will be evaluated 1 month after botulinum toxin injection.
  muscle tone 0 (0) - No increase in muscle tone 1 (1) - Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension
  1+ (2) - Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM 2 (3) - More marked increase in muscle tone through most of the ROM, but affect part(s) easily moved 3 (4) - Considerable increase in muscle tone passive, movement difficult 4 (5) - Affected part(s) rigid in flexion or extension
Modified Ashworth Scale | T3:Patients will be evaluated 3 months after botulinum toxin injection.
  muscle tone 0 (0) - No increase in muscle tone 1 (1) - Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension
  1+ (2) - Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM 2 (3) - More marked increase in muscle tone through most of the ROM, but affect part(s) easily moved 3 (4) - Considerable increase in muscle tone passive, movement difficult 4 (5) - Affected part(s) rigid in flexion or extension
Modified Ashworth Scale | T4:Patients will be evaluated 6 months after botulinum toxin injection.
  muscle tone 0 (0) - No increase in muscle tone 1 (1) - Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension
  1+ (2) - Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM 2 (3) - More marked increase in muscle tone through most of the ROM, but affect part(s) easily moved 3 (4) - Considerable increase in muscle tone passive, movement difficult 4 (5) - Affected part(s) rigid in flexion or extension
Range of Motion | T0:Patients will be evaluated before botulinum toxin injection.
  The joint is positioned according to the anatomical position and this position is considered as 0 starting position. Active and passive joint movement is measured with the help of a goniometer.
Range of Motion | T1:Patients will be evaluated 1 week after botulinum toxin injection.
  The joint is positioned according to the anatomical position and this position is considered as 0 starting position. Active and passive joint movement is measured with the help of a goniometer.
Range of Motion | T2:Patients will be evaluated 1 month after botulinum toxin injection.
  The joint is positioned according to the anatomical position and this position is considered as 0 starting position. Active and passive joint movement is measured with the help of a goniometer.
Range of Motion | T3:Patients will be evaluated 3 months after botulinum toxin injection.
  The joint is positioned according to the anatomical position and this position is considered as 0 starting position. Active and passive joint movement is measured with the help of a goniometer.
Range of Motion | T4:Patients will be evaluated 6 months after botulinum toxin injection.
  The joint is positioned according to the anatomical position and this position is considered as 0 starting position. Active and passive joint movement is measured with the help of a goniometer.
BIDA( Bodily Functioning Assessment Tool) | T0:Patients will be evaluated before botulinum toxin injection.
  The BIDA has been created to evaluate functional status, to assess therapeutic needs and changes after treatment in 2 to 18 years old children and adolescents who have orthopedic problems. The BIDAhas three forms; parent form for children, parent and self report forms for adolescents. Instrument has 86 items assessing 'upper extremity and physical function', 'transfer and basic mobility', 'sports and physical function', 'pain/comfort', 'happiness', 'global functioning' and 'expectations from treatment domains'.
BIDA( Bodily Functioning Assessment Tool) | T1:Patients will be evaluated 1 month after botulinum toxin injection.
  The BIDA has been created to evaluate functional status, to assess therapeutic needs and changes after treatment in 2 to 18 years old children and adolescents who have orthopedic problems. The BIDAhas three forms; parent form for children, parent and self report forms for adolescents. Instrument has 86 items assessing 'upper extremity and physical function', 'transfer and basic mobility', 'sports and physical function', 'pain/comfort', 'happiness', 'global functioning' and 'expectations from treatment domains'.
BIDA( Bodily Functioning Assessment Tool) | T2:Patients will be evaluated 3 months after botulinum toxin injection.
  The BIDA has been created to evaluate functional status, to assess therapeutic needs and changes after treatment in 2 to 18 years old children and adolescents who have orthopedic problems. The BIDAhas three forms; parent form for children, parent and self report forms for adolescents. Instrument has 86 items assessing 'upper extremity and physical function', 'transfer and basic mobility', 'sports and physical function', 'pain/comfort', 'happiness', 'global functioning' and 'expectations from treatment domains'.
BIDA( Bodily Functioning Assessment Tool) | T3:Patients will be evaluated 6 months after botulinum toxin injection.
  The BIDA has been created to evaluate functional status, to assess therapeutic needs and changes after treatment in 2 to 18 years old children and adolescents who have orthopedic problems. The BIDAhas three forms; parent form for children, parent and self report forms for adolescents. Instrument has 86 items assessing 'upper extremity and physical function', 'transfer and basic mobility', 'sports and physical function', 'pain/comfort', 'happiness', 'global functioning' and 'expectations from treatment domains'.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University School of Medicine Department of Physical Medicine and Rehabilitation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No